CLINICAL TRIAL: NCT01256190
Title: A Phase 2, Randomized, Single-Blind, Controlled, Comparative Efficacy and Safety and Study of Topical Fibrocaps™ and Gelatin Sponge in Surgical Hemostasis in the Netherlands
Brief Title: A Study of Fibrocaps in Liver Surgery in the Netherlands
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FC-002 NL
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Hemorrhage
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Fibrin Tissue Adhesive; Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrocaps + Gelatin sponge (Experimental): Topical Fibrocaps powder followed by application of gelatin sponge
  Interventions: Biological: Fibrocaps (fibrin sealant); Device: Gelatin sponge
- Gelatin Sponge (Active Comparator): approved device for surgical bleeding
  Interventions: Device: Gelatin sponge

INTERVENTIONS:
Biological: Fibrocaps (fibrin sealant) — human thrombin and fibrinogen topical powder
  Other Names: PRO-0601; Fibrin Sealant
  Arms: Fibrocaps + Gelatin sponge
Device: Gelatin sponge — absorbable gelatin sponge for topical use
  Other Names: Spongostan

SUMMARY:
A multi-center, prospective, randomized, single-blind, controlled, comparative efficacy and safety trial in subjects undergoing open liver resection surgery. The study will enroll 42 eligible subjects and be conducted at 4 sites in the Netherlands.

DETAILED DESCRIPTION:
This will be a multi-center, prospective, randomized, single-blind, controlled, comparative efficacy and safety trial in 60 subjects undergoing hepatic resection. Subjects will be randomized in a 2:1 ratio to Fibrocaps + Gelfoam or Gelfoam on the day of surgery.

The Fibrospray device will be used to apply Fibrocaps to the Target Bleeding Site. All investigators using the Fibrospray device will be trained on the correct and safe set-up and use of Fibrocaps and the Fibrospray device prior to participating in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Subjects who are able and willing to provide written and signed informed consent
3. Willing to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits
4. Has a life expectancy of at least one year
5. Presence of mild or moderate bleeding/oozing and control by conventional surgical techniques including but not limited to suture, ligature, and cautery is ineffective or impractical

Exclusion Criteria:

1. Pregnant or lactating women
2. Has a known intolerance to blood products or to Fibrocaps components
3. Unwilling to receive human blood products
4. Subject has a known allergy to porcine gelatin
5. Has a mental or physical condition that would, in the opinion of the Investigator, place the subject at an unacceptable risk or render the subject unable to meet the requirements of the protocol
6. Currently participating or has participated in another clinical study involving another investigational agent within 4 weeks of the planned date of surgery, or is planning participation in another clinical trial during the 4 weeks after surgery
7. Has any clinically-significant coagulation disorder that may interfere with the assessment of efficacy or pose a safety risk to the subject according to the Investigator
8. Platelets(PLT) < 100 x109 PLT/L during screening
9. Activated Partial Thromboplastin Time (aPTT) > 100 seconds during screening
10. International Normalized Ratio (INR) > 2.5 during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Frohna, MD, PhD, Study Director — Mallinckrodt
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced in December 2010 and completed in October 2011 from 5 academic medical centers in the Netherlands
Period: Overall Study
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Started | 39 | 17
Completed | 37 | 17
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge | Total
Number analyzed (Participants) | 39 | 17 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 11 | 34
  >=65 years | 16 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13) | 64 (9) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 25 | 11 | 36
Region of Enrollment [Number; unit: participants]
  Netherlands | 39 | 17 | 56

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: Time from application of treatment to cessation of bleeding
Time Frame: 0-10 minutes
Population: All subjects treated with a time to hemostasis were included in the analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 39 | 17
minutes | 2.2 (1.2) | 4.4 (3.1)
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

2. Secondary Outcome: Safety
Description: Number of participants with Adverse events and clinically significant changes/findings on labs and physical examination as well as incidence of re-operation for bleeding at the target bleeding site (TBS)
Time Frame: 28 days
Population: All subjects treated were analyzed for safety. There were 39 subjects treated with Fibrocaps and 16 treated with gelatin sponge only, since 1 gel sponge subject was randomized but not treated.
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 39 | 17
participants | 31 | 10
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; Test type: Superiority or Other; p = 0.31, t-test, 2 sided

3. Secondary Outcome: Incidence of Hemostasis at 5 Minutes
Description: Number of subjects in each group that achieved hemostasis at pre-specified times after treatment
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 39 | 17
participants | 37 | 12
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; intent-to-treat analysis; Test type: Superiority or Other; p = .022, Fisher Exact

4. Secondary Outcome: Number of Subjects Achieving Hemostasis at 3 Minutes
Time Frame: 3 minutes
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 39 | 17
participants | 30 | 9
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; intent-to treat analysis; Test type: Superiority or Other; p = 0.113, Fisher Exact

5. Secondary Outcome: Number of Patients Achieving Hemostasis at 10 Minutes
Time Frame: 10 minutes
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 39 | 17
participants | 39 | 14
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; intent-to-treat analysis; Test type: Superiority or Other; p = .025, Fisher Exact

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events (AE) were collected for 28 days post treatment
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Serious Adverse Events (participants affected / at risk) | 11/39 | 3/17
Other Adverse Events (participants affected / at risk) | 31/39 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrocaps + Gelatin Sponge (N=39) | Gelatin Sponge (N=17)
metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
peritoneal infection (Infections and infestations) | 0 (0) | 1 (1)
hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0)
post procedural bile leak (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
delirium (Psychiatric disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
edema (General disorders) | 1 (1) | 0 (0)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
congestive cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrocaps + Gelatin Sponge (N=39) | Gelatin Sponge (N=17)
Constipation (Gastrointestinal disorders) | 9 (9) | 4 (4)
potassium deficiency (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
fever (General disorders) | 4 (4) | 0 (0)
gastric retention (Gastrointestinal disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 6 (6) | 4 (5)
anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
abdonminal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
wound infection (Infections and infestations) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
low potassium (Investigations) | 0 (0) | 1 (1)
haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
neutrophil count increased (Investigations) | 1 (1) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will be part of the primary publication. Each investigator may publish on the data from subjects enrolled at their site after the initial publication has been submitted.